CLINICAL TRIAL: NCT05458895
Title: Evaluating E-Cigarette Nicotine Form, Concentration, and Flavors Among Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Theodore Wagener, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: OSU-20313; NCI-2021-06437 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-09-20; First posted 2022-07-14 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: E-cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- High concentration free-base nicotine (5%), Tobacco flavor (Experimental): Participate in vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Interventions: Other: ECIG lab session 1
- High concentration nicotine salt (5%), Tobacco flavor (Experimental): Participate in vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Interventions: Other: ECIG lab session 2
- High concentration free-base nicotine (5%), Menthol flavor (Experimental): Participate in vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Interventions: Other: ECIG lab session 3
- High concentration nicotine salt (5%), Menthol flavor (Experimental): Participate in vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Interventions: Other: ECIG lab session 4
- Low concentration free-base nicotine (1%), Tobacco flavor (Experimental): Participate in vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Interventions: Other: ECIG lab session 5
- Low concentration nicotine salt (1%), Tobacco flavor (Experimental): Participate in vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Interventions: Other: ECIG lab session 6
- Low concentration free-base nicotine (1%), Menthol flavor (Experimental): Participate in vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Interventions: Other: ECIG lab session 7
- Low concentration nicotine salt (1%), Menthol flavor (Experimental): Participate in vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Interventions: Other: ECIG lab session 8

INTERVENTIONS:
Other: ECIG lab session 1 — vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Arms: High concentration free-base nicotine (5%), Tobacco flavor
Other: ECIG lab session 2 — vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Arms: High concentration nicotine salt (5%), Tobacco flavor
Other: ECIG lab session 3 — vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Arms: High concentration free-base nicotine (5%), Menthol flavor
Other: ECIG lab session 4 — vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Arms: High concentration nicotine salt (5%), Menthol flavor
Other: ECIG lab session 5 — vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Arms: Low concentration free-base nicotine (1%), Tobacco flavor
Other: ECIG lab session 6 — vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Arms: Low concentration nicotine salt (1%), Tobacco flavor
Other: ECIG lab session 7 — vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Arms: Low concentration free-base nicotine (1%), Menthol flavor
Other: ECIG lab session 8 — vaping session with e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
  Arms: Low concentration nicotine salt (1%), Menthol flavor

SUMMARY:
This clinical trial examines the influence of nicotine form, concentration, and e-liquid flavor on youth vaping behavior, as well as the heart and lung effects associated with this behavior. Electronic cigarette (e-cig) "vaping", while being promoted as a safer alternative to conventional cigarettes, has disproportionately attracted adolescents and young adults ("youth"). This trial may help researchers understand how nicotine form, concentration, and flavor affects people's vaping behaviors and health.

DETAILED DESCRIPTION:
We will examine the influence of nicotine form and concentration, and e-liquid flavor on youth vaping behavior, nicotine uptake, abuse liability, toxicant exposure, and acute cardiovascular and pulmonary effects. Participants will complete 9 vaping sessions. Each vaping session will include a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping. During the first session, participants will use their own e-cig and e-liquid; for the following 8 sessions, participants will vape a study-provided e-cig and e-liquid.

ELIGIBILITY:
Inclusion Criteria:

* A current exclusive e-cigarette user (>= 1 vaping bout per day) for at least the past 3 months (confirmed in lab by salivary cotinine)
* 21-25 years old
* Willing to abstain from all tobacco and nicotine for at least 12 hours prior to lab sessions
* Willing to complete five, 6 hour lab visits
* Able to read and speak English
* Willing to provide informed consent

Exclusion Criteria:

* Self-reported diagnosis of lung disease including asthma, cystic fibrosis, or chronic obstructive pulmonary disease
* Unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* History of cardiac event or distress within the past 3 months
* Currently pregnant (determined using urine pregnancy test), planning to become pregnant, or breastfeeding
* Use of other tobacco products > 5 days in the past month
* Current marijuana use > 5 times per month
* Currently engaging in a vaping cessation attempt
* Ohio State University (OSU) verifies study project 2 current membership/past participation

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore L Wagener, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center; Marielle Brinkman, BS, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho YJ, Mehta T, Hinton A, Sloan R, Nshimiyimana J, Tackett AP, Roberts ME, Brinkman MC, Wagener TL. E-Cigarette Nicotine Delivery Among Young Adults by Nicotine Form, Concentration, and Flavor: A Crossover Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2426702. doi: 10.1001/jamanetworkopen.2024.26702. PMID 39120901
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Population: Full population of participants evaluated at baseline
Period: Overall Study
Arm/Group | Overall Population
Started | 88
Usual Brand e-Cigarette | 87
Low Concentration Free-base Nicotine (1%), Menthol Flavor | 65
Low Concentration Free-base Nicotine (1%), Tobacco Flavor | 64
Low Concentration Nicotine Salt (1%), Menthol Flavor | 61
Low Concentration Nicotine Salt (1%), Tobacco Flavor | 64
High Concentration Free-base Nicotine (1%), Menthol Flavor | 64
High Concentration Free-base Nicotine (1%), Tobacco Flavor | 63
High Concentration Nicotine Salt (1%), Menthol Flavor | 60
High Concentration Nicotine Salt (1%), Tobacco Flavor | 65
Completed | 60
Not Completed | 28
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 17
Not completed — Pregnancy | 2
Not completed — Withdrawal by Study Team | 1

BASELINE CHARACTERISTICS:
Population: Demographics are presented as a whole for this cross-over study and not by product order due to the large number of product orderings used to randomize the presentation order of the 8 different products.
Arm/Group | Overall Population
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.36 (1.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 73
  More than one race | 1
  Unknown or Not Reported | 1
Years of regular e-cigarette use [Mean (Standard Deviation); unit: years] — Population: Two participants failed to provide the age at which they began regularly using e-cigarettes
  years
    number analyzed (Participants) | 85
    (all) | 3.29 (2.13)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Nicotine Concentration
Description: Plasma nicotine concentration from blood drawn (3mL) 4 times in each session at baseline (0 min), 5 min., 10 min., 35 min.
Time Frame: 0, 5, 10, 35 min.
Population: Number analyzed is slightly different at each of the time points due to missing blood draws
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- Low Concentration Free-base Nicotine (1%), Menthol Flavor: Participate in vaping session with menthol flavored low concentration free-base nicotine (1%) e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
- Low Concentration Free-base Nicotine (1%), Tobacco Flavor: Participate in vaping session with tobacco flavored low concentration free-base nicotine (1%) e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
- Low Concentration Nicotine Salt (1%), Menthol Flavor: Participate in vaping session with menthol flavored low concentration nicotine salt (1%) e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
- Low Concentration Nicotine Salt (1%), Tobacco Flavor: Participate in vaping session with tobacco flavored low concentration nicotine salt (1%) e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
- High Concentration Free-base Nicotine (5%), Menthol Flavor: Participate in vaping session with menthol flavored high concentration free-base nicotine (5%) e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
- High Concentration Free-base Nicotine (5%), Tobacco Flavor: Participate in vaping session with tobacco flavored high concentration free-base nicotine (5%) e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
- High Concentration Nicotine Salt (5%), Menthol Flavor: Participate in vaping session with menthol flavored high concentration nicotine salt (5%) e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
- High Concentration Nicotine Salt (5%), Tobacco Flavor: Participate in vaping session with tobacco flavored high concentration nicotine salt (5%) e-liquid including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
- Usual Brand: Participate in vaping session with their usual brand e-cigarette including a standardized, 5-minute, 10-puff vaping bout (30 seconds between each puff) followed by 30 minutes of ad libitum (as desired) vaping.
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor | Usual Brand
Number analyzed (Participants) | 63 | 60 | 60 | 63 | 62 | 62 | 59 | 62 | 83
ng/ml
  Baseline | 0.78 [0.32 to 1.65] | 1.08 [0.45 to 2.34] | 0.89 [0.35 to 1.89] | 1.16 [0.49 to 2.62] | 0.80 [0.30 to 1.92] | 0.88 [0.38 to 2.10] | 1.03 [0.48 to 2.36] | 1.01 [0.51 to 2.21] | 0.43 [0.19 to 0.83]
  5 Minutes: number analyzed (Participants) | 62 | 58 | 57 | 61 | 58 | 60 | 56 | 62 | 77
  5 Minutes | 3.04 [1.59 to 5.16] | 2.63 [1.32 to 4.73] | 4.47 [2.30 to 7.61] | 4.66 [2.61 to 8.10] | 3.63 [1.72 to 6.15] | 3.29 [1.68 to 5.80] | 7.83 [4.33 to 16.90] | 8.76 [4.13 to 14.90] | 12.50 [7.49 to 19.30]
  10 Minutes: number analyzed (Participants) | 61 | 57 | 56 | 60 | 58 | 58 | 55 | 59 | 77
  10 Minutes | 3.12 [2.02 to 5.76] | 3.18 [1.75 to 5.17] | 4.92 [2.35 to 7.07] | 4.66 [2.67 to 7.27] | 4.45 [2.46 to 7.90] | 4.14 [1.81 to 7.18] | 8.10 [4.97 to 19.10] | 7.02 [4.29 to 16.60] | 14.10 [8.11 to 21.00]
  35 Minutes: number analyzed (Participants) | 61 | 59 | 57 | 60 | 60 | 59 | 55 | 61 | 80
  35 Minutes | 4.46 [2.45 to 8.35] | 3.51 [2.07 to 7.44] | 5.97 [2.91 to 10.70] | 5.28 [2.98 to 11.45] | 6.39 [3.59 to 13.95] | 4.23 [2.19 to 10.70] | 12.90 [6.00 to 27.30] | 10.60 [4.47 to 21.60] | 20.40 [10.25 to 31.60]

2. Primary Outcome: Puff Count
Description: E-cig puff topography data collection for abuse liability. Number of puffs taken during the 30 minutes of ad libitum (as desired) vaping session.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: Number of Puffs
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor | Usual Brand
Number analyzed (Participants) | 65 | 64 | 61 | 64 | 64 | 63 | 60 | 65 | 87
Number of Puffs | 16.17 (12.04) | 16.67 (13.84) | 17.67 (13.54) | 17.88 (13.90) | 12.52 (12.13) | 11.29 (12.64) | 14.50 (11.80) | 13.97 (12.07) | 12.40 (10.69)

3. Primary Outcome: Average Puff Duration
Description: E-cig puff topography data collection for abuse liability. Average puff duration during the 30 minutes of ad libitum (as desired) vaping session, in seconds.
Time Frame: 30 minutes
Population: Participants who attended the study visit and whose puff duration was able to be recorded.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Puffs
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor | Usual Brand
Number analyzed (Participants) | 56 | 55 | 57 | 58 | 46 | 41 | 55 | 54 | 77
Number analyzed (Puffs) | 1051 | 1067 | 1078 | 1144 | 801 | 711 | 870 | 908 | 1079
seconds | 3.20 (1.04) | 3.04 (1.08) | 3.16 (1.07) | 3.15 (1.10) | 2.65 (0.92) | 2.57 (0.97) | 2.77 (1.03) | 2.75 (1.08) | 2.70 (1.15)

4. Primary Outcome: Average Puff Volume
Description: E-cig puff topography data collection for abuse liability. The total volume of all puffs taken for each participant during the 30 minutes of ad libitum (as desired) vaping session, in ml.
Time Frame: 30 minutes
Population: Participants who attended the study visit and whose puff volume was able to be recorded.
Measure: Mean (Standard Deviation); unit: ml
Units Other Than Participants: Puffs
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor | Usual Brand
Number analyzed (Participants) | 64 | 62 | 59 | 61 | 53 | 54 | 57 | 58 | 82
Number analyzed (Puffs) | 1051 | 1067 | 1078 | 1144 | 801 | 711 | 870 | 908 | 1079
ml | 48.68 (17.28) | 46.31 (18.44) | 50.64 (22.05) | 51.92 (30.01) | 36.82 (12.13) | 35.12 (13.16) | 41.76 (15.35) | 40.86 (17.26) | 69.29 (40.42)

5. Primary Outcome: Lung Function Assessment
Description: Lung function data will be collect using a handheld spirometry device. Physiological effects of pulmonary function collected from inhaled and exhaled breaths. Measures amount inhaled and how quickly exhaled.
  Change from baseline in forced expiratory volume (FEV) Change from baseline in forced vital capacity (FVC)
Time Frame: Baseline and 35 minutes
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor | Usual Brand
Number analyzed (Participants) | 65 | 64 | 61 | 64 | 64 | 63 | 60 | 65 | 87
Liters
  FEV | -0.03 (0.21) | -0.05 (0.21) | -0.01 (0.19) | 0.003 (0.24) | -0.08 (0.40) | -0.02 (0.38) | -0.05 (0.24) | -0.04 (0.24) | 0.09 (0.39)
  FVC | -0.02 (0.29) | -0.01 (0.25) | -0.0006 (0.24) | 0.30 (2.36) | -0.12 (0.53) | -0.02 (0.53) | -0.01 (0.37) | -0.23 (1.68) | 0.13 (0.42)

6. Primary Outcome: Airway Inflammation (NIOX VERO)
Description: Physiological effects of pulmonary function collected from inhaled and exhaled breaths. Airway inflammation will be assessed using exhaled nitric oxide via the NIOX VERO.
Time Frame: 35 minutes
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor | Usual Brand
Number analyzed (Participants) | 65 | 64 | 61 | 64 | 64 | 63 | 60 | 65 | 87
ppb | 18.94 (11.52) | 19.27 (13.38) | 18.95 (12.14) | 19.69 (11.86) | 18.52 (12.76) | 21.94 (19.51) | 19.20 (11.43) | 20.02 (12.55) | 18.77 (12.70)

7. Secondary Outcome: Sensory E-Cigarette Expectancies Scale (SEES)
Description: Background measures. Comprised of 9 items each of which range 0-4 from "never" to "almost always".
  The 3 subscales (enjoyment of taste and smell, pleasurable physical sensations, enjoyment of vapor cloud production) are the average of 3 items each; scores range from 0 to 4 with higher scores indicating greater enjoyment.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 87
score on a scale
  Enjoyment of Taste and Smell | 2.69 (0.77)
  Pleasurable Physical Sensations | 2.76 (0.87)
  Enjoyment of Vapor Cloud Production | 1.66 (1.06)

8. Secondary Outcome: Modified Cigarette Dependence Scale
Description: Assess e-cigarette dependence.
  Scores range from 5 to 25 with higher scores indicating a greater level of dependence.
Time Frame: Baseline
Population: Participants who responded to all items on the modified cigarette dependence scale at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 83
score on a scale | 17.37 (4.18)

9. Secondary Outcome: Drug Effects/Liking Questionnaire
Description: An adapted version of the Drug Effects/Liking Questionnaire will assess the desire and liking of UBMC and all three study products, positive and negative effects (i.e., side effects), and perceived strength and effectiveness. Five visual analog scale items ranging from 0 ('not at all') to 100 ('extremely') assessed wanting to smoke the product again, liking the product, enjoying the product, finding the product pleasurable and satisfying.
Time Frame: 35 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor | Usual Brand
Number analyzed (Participants) | 65 | 64 | 61 | 64 | 64 | 63 | 60 | 65 | 87
score on a scale
  Want | 40.40 (23.83) | 32.59 (23.08) | 44.69 (26.44) | 37.78 (22.14) | 27.48 (25.41) | 17.16 (21.13) | 43.58 (24.87) | 29.75 (24.76) | 45.40 (20.93)
  Like | 47.54 (25.32) | 35.36 (25.34) | 48.82 (27.28) | 41.94 (24.30) | 27.44 (27.40) | 17.08 (21.59) | 49.67 (27.13) | 31.51 (25.04) | 69.05 (21.81)
  Enjoy | 46.51 (25.12) | 36.70 (26.42) | 49.66 (27.01) | 43.02 (25.03) | 27.39 (26.77) | 18.27 (21.24) | 50.02 (25.74) | 31.42 (25.05) | 72.57 (17.73)
  Pleasurable | 46.28 (24.26) | 36.42 (24.96) | 50.23 (26.53) | 44.66 (23.63) | 29.33 (27.92) | 18.60 (20.17) | 52.13 (25.00) | 34.48 (24.97) | 72.57 (15.94)
  Satisfying | 44.89 (24.35) | 37.45 (23.26) | 48.84 (26.06) | 41.98 (25.56) | 33.95 (26.97) | 25.05 (23.64) | 52.48 (23.69) | 39.69 (26.24) | 74.33 (15.34)

10. Secondary Outcome: Modified Cigarette Evaluation Questionnaire (mCEQ)
Description: The modified Cigarette Evaluation Questionnaire (mCEQ) will assess subjective responses to e-cigarettes (e.g., reward, satisfaction). The 12-item mCEQ includes five subscales: Smoking Satisfaction, Psychological Reward, Aversion, Enjoyment of Respiratory Tract Sensations, and Craving Reduction, with items rated from 1 (not at all) to 7 (extremely likely). Items are averaged to create each of the subscales also ranging from 1 to 7 with higher values indicating greater levels of smoking satisfaction, psychological reward, aversion, enjoyment of respiratory tract sensations, an craving reduction.
Time Frame: 35 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor
Number analyzed (Participants) | 65 | 64 | 61 | 64 | 64 | 63 | 60 | 65
score on a scale
  Satisfaction | 3.35 (1.32) | 2.78 (1.04) | 3.58 (1.31) | 2.97 (1.07) | 2.93 (1.33) | 2.26 (0.97) | 3.80 (1.39) | 2.93 (1.22)
  Reward | 2.19 (0.99) | 2.17 (0.81) | 2.35 (1.10) | 2.23 (0.98) | 2.24 (1.13) | 2.01 (0.94) | 2.50 (1.18) | 2.32 (1.16)
  Aversion | 1.18 (0.43) | 1.31 (0.57) | 1.29 (0.50) | 1.35 (0.95) | 1.63 (0.86) | 1.63 (0.74) | 1.73 (1.10) | 1.78 (1.25)
  Sensation | 3.20 (1.55) | 2.55 (1.30) | 3.62 (1.66) | 2.83 (1.34) | 2.22 (1.50) | 1.73 (1.19) | 3.32 (1.57) | 2.77 (1.48)
  Craving | 3.25 (1.58) | 3.17 (1.44) | 3.39 (1.38) | 3.23 (1.44) | 3.45 (1.58) | 2.97 (1.54) | 4.05 (1.68) | 3.40 (1.53)

11. Secondary Outcome: E-cigarette Purchase Task - Breakpoint
Description: Behavioral economic demand Asks participants how much they would be willing to pay (ranging from 0¢ to $1,120) for a puff of their study product. Specifically they will be asked, "Thinking about the study product, how many puffs of e-cigarette would you smoke if they were each at the following prices?". Breakpoint is the first price of zero consumption.
Time Frame: 35 minutes
Measure: Median (Inter-Quartile Range); unit: Dollars
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor | Usual Brand
Number analyzed (Participants) | 65 | 64 | 61 | 64 | 64 | 63 | 60 | 65 | 86
Dollars | 0.5 [0.25 to 2] | 0.38 [0.05 to 2.5] | 1 [0.25 to 3] | 0.5 [0.25 to 3] | 0.5 [0.13 to 4] | 0.25 [0 to 2] | 1 [0.25 to 3.5] | 0.5 [0.13 to 2] | 2.0 [0.5 to 6.0]

12. Secondary Outcome: Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form
Description: E-cig craving/suppression of craving and withdraw will be measured using the Tiffany-Drobes Questionnaire of Smoking Urges (QSU): Brief Form with a modified version (replacing the word "cigarette" with "e-cigarette"). This is a 10-item measure where participants rate smoking/vaping-related items on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Similar to previous studies, we will collapse the items into two previously identified factors (Factor 1: strong desire and intention to smoke/vape; Factor 2: anticipation of relief from withdrawal symptoms). Scores are calculated by summing the items and range from 5 to 35 for each of the factors with higher scores indicating greater craving to smoke/vape.
Time Frame: 0, 5, 10, 35 min.
Population: Participants who attended the study product visit and fully completed the QSU items
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor | Usual Brand
Number analyzed (Participants) | 65 | 64 | 61 | 64 | 64 | 63 | 60 | 65 | 87
units on a scale
  QSU Desire: 0min | 24.85 (8.27) | 25.44 (7.02) | 25.51 (7.43) | 25.56 (7.15) | 24.52 (7.26) | 25.25 (7.55) | 24.03 (7.85) | 24.09 (7.97) | 26.18 (7.44)
  QSU Relief: 0min | 13.78 (7.18) | 13.88 (7.02) | 14.28 (7.18) | 14.08 (7.22) | 13.69 (7.14) | 13.68 (6.83) | 13.25 (7.35) | 13.80 (7.74) | 15.64 (6.92)
  QSU Desire: 5 min: number analyzed (Participants) | 65 | 64 | 61 | 64 | 64 | 63 | 60 | 65 | 85
  QSU Desire: 5 min | 18.92 (7.63) | 18.38 (6.78) | 19.54 (7.43) | 19.00 (7.50) | 16.34 (7.47) | 17.44 (7.74) | 16.78 (7.02) | 16.98 (7.13) | 14.45 (6.85)
  QSU Relief: 5min | 10.77 (6.14) | 10.56 (5.40) | 10.98 (5.82) | 10.77 (5.39) | 10.08 (5.58) | 10.35 (5.91) | 9.95 (5.40) | 10.02 (4.97) | 9.95 (4.84)
  QSU Desire: 10 min | 17.49 (8.04) | 17.22 (6.96) | 17.64 (7.54) | 17.73 (7.46) | 15.29 (7.11) | 16.56 (7.56) | 15.15 (6.88) | 15.74 (6.83) | 13.76 (6.75)
  QSU Relief: 10 min | 9.92 (5.82) | 10.03 (4.97) | 9.93 (5.44) | 9.92 (5.13) | 9.23 (4.71) | 9.71 (5.30) | 9.37 (4.96) | 9.66 (4.84) | 9.40 (5.05)
  QSU Desire: 35 min | 16.17 (7.94) | 16.72 (7.68) | 16.87 (7.02) | 16.88 (7.79) | 15.41 (7.15) | 16.54 (7.65) | 14.55 (6.45) | 14.92 (7.48) | 12.49 (5.83)
  QSU Relief: 35 min | 9.57 (5.51) | 9.58 (4.63) | 9.41 (4.68) | 9.28 (4.53) | 8.94 (4.56) | 9.38 (4.45) | 8.40 (3.82) | 8.95 (4.55) | 8.09 (4.29)

13. Secondary Outcome: Vascular Reactivity
Description: Endothelial function will be collected through EndoPAT device. Specifically, the natural log of RHI, the reactive hyperemia index, will be recorded.
  The RHI (Reactive Hyperemia Index) or LnRHI (natural log of RHI) is the post-to-pre occlusion PAT™ signal ratio in the occluded arm, relative to the same ratio in the control arm, corrected for baseline vascular tone. Values less than 1.67 or higher than 0.51 are considered to be abnormal.
Time Frame: Pre-Vaping Session at Visit 1
Population: Participants who attended the baseline study visit and whose endothelial function was able to be recorded with the EndoPAT device.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Overall Population: All participants included in the study
Arm/Group | Overall Population
Number analyzed (Participants) | 86
ratio | 0.47 (0.26)

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Low Concentration Free-base Nicotine (1%), Menthol Flavor | Low Concentration Free-base Nicotine (1%), Tobacco Flavor | Low Concentration Nicotine Salt (1%), Menthol Flavor | Low Concentration Nicotine Salt (1%), Tobacco Flavor | High Concentration Free-base Nicotine (5%), Menthol Flavor | High Concentration Free-base Nicotine (5%), Tobacco Flavor | High Concentration Nicotine Salt (5%), Menthol Flavor | High Concentration Nicotine Salt (5%), Tobacco Flavor | Usual Brand
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/64 | 0/61 | 0/64 | 0/64 | 0/63 | 0/60 | 0/65 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/64 | 0/61 | 0/64 | 0/64 | 0/63 | 0/60 | 0/65 | 0/87
Other Adverse Events (participants affected / at risk) | 0/65 | 0/64 | 0/61 | 0/64 | 0/64 | 0/63 | 0/60 | 0/65 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT05458895/Prot_SAP_ICF_000.pdf